CLINICAL TRIAL: NCT02145728
Title: The Effect of Cognitive Functional Therapy on Patients With Non-specific Chronic Low Back Pain: a Multi-centre Randomized Trial
Brief Title: The Effect of Cognitive Functional Therapy on Patients With Non-specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Curtin University (Other); KU Leuven (Other); Mayo General Hospital, Ireland (Other); Health Service Executive, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGH-14-UL
Record Dates: First submitted 2014-04-30; First posted 2014-05-23 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Chronic Low Back Pain
Keywords: Non-specific chronic low back pain; Cognitive functional therapy; Exercise classes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Cognitive Functional Therapy (Experimental): The intervention being tested has four main components: (1) a cognitive component, for each patient, their vicious cycle of pain will outlined in a diagram based on their findings from the examination and the Orebro Musculoskeletal Pain Screening Questionnaire; (2) specific movement exercises designed to normalize maladaptive movement behaviours; (3) targeted functional integration of activities in their daily life previously, reported to be avoided or provocative by the patient; and (4) a physical activity and lifestyle programme.
  Interventions: Behavioral: Individual Cognitive Functional Therapy
- Group Exercise Classes (Active Comparator): 6 classes will take place in total. The class has 3 components each week. First, a 30 minute talk and discussion on chronic pain, and some tips for participants. Second, a 40 minute exercise circuit, involving aerobic exercise, and gentle stretching and strengthening exercises. Finally, a 5 minute relaxation/mindfulness session will take place at the end. The total time involved is approximately 1 hour and 15 minutes.
  Interventions: Behavioral: Group Exercise Classes

INTERVENTIONS:
Behavioral: Individual Cognitive Functional Therapy — Cognitive functional therapy (CFT) is a novel, patient centred behavioural intervention which addresses multiple dimensions in non-specific chronic low back pain (NSCLBP). It combines a functional behavioural approach of normalising provocative postures and movements while discouraging pain behaviours, with cognitive restructuring of the NSCLBP problem.
  Arms: Individual Cognitive Functional Therapy
Behavioral: Group Exercise Classes — Each class involves a combination of education, exercise and relaxation/mindfulness. The education topics include pain and the nervous system, posture and ergonomics, exercise and relaxation and sleep. The exercise component includes 10 stations of a combination of aerobic, strength and flexibility exercises. These will be walking/jogging on the spot, mini-squats, sit to stands, wall push ups, bridging, step-ups and a combination of leg and low back stretches. The relaxation/mindfulness component will take place at the end of each class and will involve breathing and relaxation of the body.
  Arms: Group Exercise Classes

SUMMARY:
The purpose of this study is to evaluate whether individual cognitive functional therapy (CFT), when compared to group exercise classes is effective in reducing pain and disability in patients with non-specific chronic low back pain.

DETAILED DESCRIPTION:
A multi-centre randomised study with 6 month, 12 month and 36 month follow up will be used. Patient with non- specific chronic low back pain will be assessed for eligibility. The patients fitting the inclusion criteria will be randomised to receive either the individual CFT or the group classes consisting of education and exercise. Participants' pain, disability, socio-economic status, beliefs, fear, catastrophizing, self-efficacy, general health, stress levels, as well as number and cost of treatments will be evaluated using a range of outcome measures at the start and on completion of the treatment. Patients will receive another copy of the questionnaires in the post at 6 month, 12 months and 36 months after treatment to reassess clinical outcomes. If a participant does not respond to follow-up, they will be telephoned to ask if they wish to complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75
* Chronic low back pain greater than 6 months duration
* Score greater than 14% for disability on Oswestry Disability Index (ODI)
* Independently mobile (with or without aids), to be capable of participating in a rehabilitation programme

Exclusion Criteria:

* Primary pain area is not the lumbar spine (from T12-buttocks)
* Leg pain as the primary problem (nerve root compression or disc prolapse with true radicular pain/radiculopathy, lateral recess/central or spinal stenosis with primary leg pain)
* <6 months post lumbar spine or lower limb or abdominal surgery
* Pain relieving procedures such as injection based therapy (e.g epidurals) and day case procedures (e.g rhizotomy) in the last 3 months
* Pregnancy
* Rheumatologic/inflammatory disease (e.g. rheumatoid arthritis (RA), ankylosing spondylitis (AS), psoriatic arthritis, lupus, scheuermann's disease)
* Progressive neurological disease (e.g. multiple sclerosis (MS), parkinson's disease (PD), motor neuron disease (MND)
* Unstable cardiac conditions
* Red flag disorders like malignancy/cancer, acute traumas like fracture (<6 months ago) or infection, spinal cord compression/cauda equina

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Used to assess change in disability levels over the course of the trial and follow-up

SECONDARY OUTCOMES:
Numerical rating scale (NRS) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Measures pain intensity
Socio-economic Conditions Index | Baseline
  Measures socio-economic status
Back Pain Beliefs Questionnaire | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assess a person's beliefs about their back pain
Physical activity subscale of the Fear-Avoidance Beliefs Questionnaire (FABQ) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assesses a person's level of fear-avoidance beliefs regarding physical activities.
The catastrophising subscale of the Coping Strategies Questionnaire (CSQ) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assesses level of pain catastrophizing.
Pain Self- Efficacy Questionnaire (PSEQ) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assesses level of pain self-efficacy
Subjective Health Complaints Inventory (SHC) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assess level of subjective health complaints
Nordic Musculoskeletal Screening Questionnaire | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assesses areas of bodily pain
Stress subscale of the Depression, Anxiety and Stress scale (DASS 21) | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  Assesses patient's stress levels.
Patient Satisfaction Questionnaire | At 8-14 weeks
  Assesses patient satisfaction
Short-Form Orebro Musculoskeletal Screening Questionnaire (OMSQ) | Measured at baseline
  Stratifies patients into low, medium or high risk of delayed pain recovery and chronicity.
Medication usage | Baseline, post intervention (at 8-14 weeks), 6, 12 and 36 months
  To assess changes in levels of medication used.
Economic evaluation | 6, 12 and 36 months
  Assesses direct and indirect costs of both treatment arms to see which is more cost-effective.
Level of co-interventions | Baseline, post-intervention (at 8-14 weeks), 6, 12 and 36 months
  Assesses the number/type of healthcare services availed of throughout the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kieran O' Sullivan, PhD, Study Director — University of Limerick; Mary O'Keeffe, BSc Physio, Principal Investigator — University of Limerick; Prof. Peter O'Sullivan, Professor, Principal Investigator — Curtin University; Dr Norelee Kennedy, PhD, Principal Investigator — University of Limerick; Prof. Wim Dankaerts, Professor, Principal Investigator — KU Leuven
Locations (3):
- Ireland (3):
  - Ballina Primary Care Centre, Mayo, Connacht
  - Claremorris Primary Care Centre, Mayo, Connacht
  - Mayo General Hospital, Mayo, Connacht

REFERENCES:
- [Background] O'Sullivan P. It's time for change with the management of non-specific chronic low back pain. Br J Sports Med. 2012 Mar;46(4):224-7. doi: 10.1136/bjsm.2010.081638. Epub 2011 Aug 4. No abstract available. PMID 21821612
- [Result] Vibe Fersum K, O'Sullivan P, Skouen JS, Smith A, Kvale A. Efficacy of classification-based cognitive functional therapy in patients with non-specific chronic low back pain: a randomized controlled trial. Eur J Pain. 2013 Jul;17(6):916-28. doi: 10.1002/j.1532-2149.2012.00252.x. Epub 2012 Dec 4. PMID 23208945
- [Derived] O'Keeffe M, O'Sullivan P, Purtill H, Bargary N, O'Sullivan K. Cognitive functional therapy compared with a group-based exercise and education intervention for chronic low back pain: a multicentre randomised controlled trial (RCT). Br J Sports Med. 2020 Jul;54(13):782-789. doi: 10.1136/bjsports-2019-100780. Epub 2019 Oct 19. PMID 31630089
- [Derived] O'Keeffe M, Purtill H, Kennedy N, O'Sullivan P, Dankaerts W, Tighe A, Allworthy L, Dolan L, Bargary N, O'Sullivan K. Individualised cognitive functional therapy compared with a combined exercise and pain education class for patients with non-specific chronic low back pain: study protocol for a multicentre randomised controlled trial. BMJ Open. 2015 Jun 1;5(6):e007156. doi: 10.1136/bmjopen-2014-007156. PMID 26033941